CLINICAL TRIAL: NCT05826483
Title: Exploration of the Clinical Application of Almonertinib in the First-line Treatment of Patients With EGFR Mutation-positive Advanced Non-small Cell Lung Cancer With Poor Performance Status
Brief Title: Almonertinib in the First-line Treatment of Patients of NSCLC With Poor Performance Status
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Zhou Chengzhi, Director, Head of pneumology department, Principal Investigator, Clinical Professor, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROC202201
Record Dates: First submitted 2022-02-05; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Malignant Tumor of Lung; Poor Performance Status
Keywords: Almonertinib; Non-Small Cells Lung Cancer; poor performance status
MeSH Terms: conditions — Lung Neoplasms | interventions — aumolertinib

STUDY DESIGN:
Intervention Model Description: Single Group Assignment Almonertinib monotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Almonertinib (Experimental): Almonertinib, 110 mg, po, QD; 28 days every cycle
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — Almonertinib Mesilate Tablets

SUMMARY:
Most of the lung cancer patients treated in hospitals in China are in advanced stage, accounting for more than 2/3 of all lung cancer patients, and some of the patients have a poor performence status.At present, most of the patients included in clinical trials are patients with good PS score, and the NCCN guidelines for advanced lung cancer patients with poor performence status recommend the best supportive care.Therefore, the investigator wanted to explore the efficacy and safety of Almonertinib in lung cancer patients with poor performance status.

DETAILED DESCRIPTION:
Most of the lung cancer patients treated in hospitals in China are in advanced stage, accounting for more than 2/3 of all lung cancer patients, and some of the patients have a poor performence status.In recent years, systemic treatments with good efficacy and low toxicity, such as gene-targeted therapy, anti-angiogenic therapy and immunotherapy, have largely replaced single chemotherapy, and have great potential to benefit from existing treatments for poor PS scores of advanced lung cancer patients can adopt more aggressive treatment strategies.At present, most of the patients included in clinical trials are patients with good PS score, and the NCCN guidelines for advanced lung cancer patients with poor performence status recommend the best supportive care.Therefore,the investigator wanted to explore the efficacy and safety of Almonertinib in lung cancer patients with poor performance status.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up.
2. Male or female who is over 18 years old.
3. Malignant tumorsr proved by pathology.
4. NSCLC patients with EGFR mutation (19 deletion/21 L858R point mutation) or primary T790M mutation in pre-enrollment genetic testing.
5. PS score of 2-4; this score is caused by complications caused by the tumor and cannot be improved by any non-anti-tumor means.
6. Patients with brain metastases may be enrolled at the discretion of the investigator.
7. Appropriate organ system function.

Exclusion Criteria:

1. Patients who have previously used any antineoplastic drugs。
2. Small cell lung cancer (including lung cancer mixed with small cell lung cancer and non-small cell lung cancer);
3. Genetic testing results in patients with rare EGFR genotypes (G719X, E709X, Del18 on exon 18, Ins19 on exon 19, Ins20, S768I on exon 20, and L861Q on exon 21).
4. Patients with other mutations (ALK, Ros-1, C-MET).
5. Imperfection of upper gastrointestinal physiology, or absorption disorder syndrome, or inability to tolerate oral drugs, or active peptic ulcer;
6. Participated in other clinical trials within 4 weeks before the start of the study;
7. patients with hypertension who cannot control well through single antihypertensive medication (systolic blood pressure > 140mmhg, diastolic blood pressure > 90mmhg), myocardial ischemia or myocardial infarction, arrhythmia (including QT interval > 440 ms) or cardiac insufficiency;
8. Allergic to any ingredient in the drug;
9. Patients with abnormal coagulation function, receiving thrombolysis or anticoagulation therapy, bleeding tendency or have clear gastrointestinal bleeding concerns;
10. Hyperactive/venous thrombosis events, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism occurred in 6 months before the start of the study;
11. Wound or fracture has not been healed for a long time;
12. urinary protein was greater than ++ and 24-hour urinary protein quantification #1.0 g.
13. Severe or uncontrolled infections;
14. Substance abuse or mental disorder;
15. Objective evidence of a history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radioactive pneumonia, drug-related pneumonia, and severe impairment of pulmonary function;
16. Immunodeficiency, including being HIV-positive, or having other acquired, congenital immunodeficiency diseases, or having a history of organ transplantation;
17. Other malignant tumors within 5 years, except cured basal cell carcinoma of the skin and orthotopic carcinoma of the cervix;
18. Who have received VEGFR inhibitors, such as sorafenib and sunitinib, etc.;
19. pregnant or lactating women;
20. the researchers considered it unsuitable for inclusion。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  Objective Response Rate
Time of PS score change from 2~4 to 1 | 6 months
  Time of performance status score change from 2~4 to 1

SECONDARY OUTCOMES:
PFS | 24 months
  Median progression-free survival
OS | from baseline until death due to any cause, up to a maximum of approximately 4years
  Median overall survival
DCR | 24 months
  Disease control rate

OTHER OUTCOMES:
Safety: Dose-limiting toxicities | from the screening period to 28 days after treatment completion
  Any level 3 or greater toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Chengzhi, MD, Study Director — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Zhou Chengzhi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
no plan